CLINICAL TRIAL: NCT00001373
Title: An Exploratory Study of the Genetics, Pathophysiology, and Natural History of Autoinflammatory Diseases
Brief Title: Familial Mediterranean Fever and Related Disorders: Genetics and Disease Characteristics
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: University of Massachusetts, Worcester (Other); Duke University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940105; 94-HG-0105
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-20

CONDITIONS: Familial Mediterranean Fever (FMF); Autoinflammation; Periodic Fever; Fever; Genetic Diseases; ROSAH; ALPK1
Keywords: Splenomegaly; Retinal Dystrophy; Periodic Fever; Optic Nerve Edema; HEADACHE; Genetics; Familial Mediterranean; Autoinflammation; Anhidrosis; Alpha-Kinase 1
MeSH Terms: conditions — Familial Mediterranean Fever; Hereditary Autoinflammatory Diseases; Fever; Genetic Diseases, Inborn; Splenomegaly; Retinal Dystrophies; Headache; Hypohidrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected: Patients with auto-inflammatory disorders
- Family Members: Family members of patients
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
This study is designed to explore the genetics and pathophysiology of diseases presenting with intermittent fever, including familial Mediterranean fever, TRAPS, hyper-IgD syndrome, and related diseases.

The following individuals may be eligible for this natural history study: 1) patients with known or suspected familial Mediterranean fever, TRAPS, hyper-IgD syndrome or related disorders; 2) relatives of these patients; 3) healthy, normal volunteers 7 years of age or older.

Patients will undergo a medical and family history, physical examination, blood and urine tests. Additional tests and procedures may include the following:

1. X-rays
2. Consultations with specialists
3. DNA sample collection (blood or saliva sample) for genetic studies. These might include studies of specific genes, or more complete sequencing of the genome.
4. Additional blood samples a maximum of 1 pint (450 ml) during a 6-week period for studies of white cell adhesion (stickiness)
5. Leukapheresis for collecting larger amounts of white cells for study. For this procedure, whole blood is collected through a needle in an arm vein. The blood flows through a machine that separates it into its components. The white cells are removed and the rest of the blood is returned to the body through another needle in the other arm.

Patients may be followed approximately every 6 months to monitor symptoms, adjust medicine dosages, and undergo routine blood and urine tests. They will receive genetic counseling by the study team on the risk of having affected children and be advised of treatment options.

Participating relatives will undergo a medical and family history, possibly with a review of medical records, physical examination, blood and urine tests. Additional procedures may include a 24-hour urine collection, X-rays, and consultations with medical specialists. A DNA sample (blood or saliva) will also be collected for genetic studies. Additional blood samples of no more than 550 mL during an 8-week period may be requested for studies of white cell adhesion (stickiness).

Relatives who have familial Mediterranean fever, TRAPS, or hyper-IgD syndrome will receive the same follow-up and counseling as described for patients above.

Normal volunteers and patients with gout will have a brief health interview and check of vital signs (blood pressure and pulse) and will provide a blood sample (up to 90 ml, or 6 tablespoons). Additional blood samples of no more than 1 pint over a 6-week period may be requested in the future.

DETAILED DESCRIPTION:
Study Description

This is an exploratory natural history protocol that will enroll patients with known or as yet undiagnosed disorders of inflammation. Blood, saliva, or buccal samples will be collected for genetic analysis, blood samples will be obtained for immunologic and other functional studies, a small number of subjects may undergo skin biopsy, leukapheresis, or bone marrow aspiration and biopsy, and some patients will be provided standard medical care follow up, with retrospective analysis of the clinical data gathered during follow up.

Objectives

Primary Objective: To discover the genetic basis of human disorders of inflammation.

Secondary Objective: To enumerate immunologic features and genotype-phenotype associations in specific inflammatory diseases.

Tertiary Objectives: To describe the clinical features of poorly characterized or newly defined disorders of inflammation, through the retrospective chart review of standard medical practice follow up and through the enrollment of selected subjects in separate, disease-specific protocols.

Endpoints

Primary Endpoints: The discovery of rare, high-penetrance genetic variants and common, low-penetrance genetic variants conferring susceptibility to inflammatory disease; the discovery of structural genomic variants (insertions, deletions, inversions, translocations, etc.) that cause human inflammatory disease; the discovery of common, low-penetrance germline variants that confer susceptibility to human inflammatory disease; and the discovery of somatic mutations that give rise to human inflammatory disease.

Secondary Endpoint: The description of immune cell populations, inflammatory mediators, gene expression profiling, epigenetic features, and ex vivo functional assays of leukocytes from subjects with specific inflammatory diseases.

Tertiary Endpoints: Given the wide range of inflammatory diseases, the endpoints will be formulated for specific conditions based on the clinical features of that condition.

ELIGIBILITY:
* INCLUSION CRITERIA:

There are three populations that will be included in this study: subjects with known or suspected autoinflammatory diseases, family members of subjects with known or suspected autoinflammatory diseases, and healthy controls. Persons interested in participation may be given a screening questionnaire to determine eligibility. Questions in the screening questionnaire are important to help us determine if subjects have known autoinflammatory diseases, or if there is a high clinical suspicion of autoinflammatory disease.

In order to be eligible to participate in this study as a subject with known or suspected autoinflammatory disease, an individual must meet all of the following criteria:

1. Stated willingness to participate in study procedures (which at the very least includes providing a mail-in sample for genetic analysis);
2. Regardless of gender, at least one month of age;
3. A medical history that, in the expert opinion of the study team, is consistent with the possibility of autoinflammatory disease; and
4. Ability of the subject, parents (in the case of children), or Legally Authorized Representative to understand and the willingness to sign a written informed consent document.

In order to be eligible to participate in this study as a family member of a subject with known or suspected autoinflammatory disease, an individual must meet all of the following criteria:

1. Stated willingness to participate in study procedures (which at the very least includes providing a mail-in sample for genetic analysis);
2. Regardless of gender, at least one month of age;
3. Relationship, either by blood or marriage, to an individual enrolled or about to be enrolled in the study with known or suspected autoinflammatory disease;
4. Likelihood, in the expert opinion of the study team, that analysis of a sample from the individual would advance genetic or functional analysis of the affected relative's possible autoinflammatory condition; and
5. Ability of the subject, parents (in the case of children), or Legally Authorized Representative to understand and the willingness to sign a written informed consent document.

In order to be eligible to participate in this study as a healthy volunteer, an individual must meet all of the following criteria:

1. Stated willingness to participate in study procedures for healthy volunteers;
2. Regardless of gender, at least one year old, and not pregnant (by history of a missed menstrual period);
3. Likelihood, in the expert opinion of the study team, that a sample from the individual would advance the functional analysis of an autoinflammatory condition under study; and
4. Ability of the subject or parents (in the case of children) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

For any of the three categories of subjects, an individual will be excluded from participation in this study if he or she has a medical condition that would, in the opinion of the investigators, confuse the interpretation of the study.

Ages: 2 Months to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoinflammatory disorders and unaffected family members, and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1994-03-10 (Actual)

PRIMARY OUTCOMES:
Genetic linkage in autoinflammatory dise | annually
  discovery of genetic associations to autoinflammatory disorders

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Solomon, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (5):
- United States (5):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Walter Reed National Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual genomic sequencing data and corresponding phenotype data will be deposited in dbGaP as part of the study's Genomic Data Sharing Plan. Non-genomic and/or phenotypic individual data will not be deposited in shared databases for broad research use.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Genomic Sharing Plan in effect since 2018 with genomic data deposited to dbGaP for broad availability within six months of final data analysis of each genomic sequence. No end date of data availability through dbGaP.
Access Criteria: Genomic sequences will be deposited to dbGaP following final sequence analysis and available for broad use, as determined by dbGaP usage committee.

REFERENCES:
- [Background] Hashkes PJ, Spalding SJ, Giannini EH, Huang B, Johnson A, Park G, Barron KS, Weisman MH, Pashinian N, Reiff AO, Samuels J, Wright DA, Kastner DL, Lovell DJ. Rilonacept for colchicine-resistant or -intolerant familial Mediterranean fever: a randomized trial. Ann Intern Med. 2012 Oct 16;157(8):533-41. doi: 10.7326/0003-4819-157-8-201210160-00003. PMID 23070486
- [Background] Aksentijevich I, Kastner DL. Genetics of monogenic autoinflammatory diseases: past successes, future challenges. Nat Rev Rheumatol. 2011 Jul 5;7(8):469-78. doi: 10.1038/nrrheum.2011.94. PMID 21727933
- [Background] Bulua AC, Mogul DB, Aksentijevich I, Singh H, He DY, Muenz LR, Ward MM, Yarboro CH, Kastner DL, Siegel RM, Hull KM. Efficacy of etanercept in the tumor necrosis factor receptor-associated periodic syndrome: a prospective, open-label, dose-escalation study. Arthritis Rheum. 2012 Mar;64(3):908-13. doi: 10.1002/art.33416. PMID 22006113
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-HG-0105.html